CLINICAL TRIAL: NCT03467620
Title: Oral Cannabidiol Capsule Usage as an Adjunct Therapy for Crohn's Disease: a Randomized, Placebo-controlled Study
Brief Title: Cannabidiol Usage as an Adjunct Therapy for Crohn's Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kyle M Geary, MD, Gastroenterology Fellow, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0529 Adm Withdrawn
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Cannabis
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Marijuana Abuse | interventions — Cannabidiol; Cannabinoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol oral capsule (Experimental): 25-mg capsule of Cannabidiol (CBD) per day taken daily for a duration of 12 weeks.
  Interventions: Drug: Cannabidiol
- Placebo oral capsule (Placebo Comparator): One placebo capsule per day for a duration of 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Cannabidiol — Administration of one oral 25-mg capsule of Cannabidiol daily for a duration of 12 weeks
  Other Names: Cannabinoid
  Arms: Cannabidiol oral capsule
Drug: Placebo oral capsule — Administration of one oral placebo capsule daily for a duration of 12 weeks
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
To date, few studies have assessed the efficacy and safety of Cannabinoids, compounds derived from the Cannabis plant, in patients with Crohn's disease. Our study seeks to pilot a randomized, placebo-controlled trial assessing the efficacy and safety of oral cannabinoids as an adjunct therapy in patients with Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease is a type of inflammatory disease which can affect any portion of the gastrointestinal tract, from the mouth to the perianal area. Symptoms depend on location of the disease, however, many patients experience some aspect of recurrent abdominal pain, nausea, emesis, and unintentional weight loss. A common and challenging dilemma is how to manage patients who continue to have some degree of symptoms despite a common treatment regimen typically consisting of corticosteroids, thiopurines, methotrexate, or anti-TNF alpha therapies. With the recent wave of medicinal cannabis legalization in many states, many patients have begun using cannabis or commercially available cannabidiol-containing compounds as an adjunct therapy for their symptoms related to chronic inflammation and pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English-speaking
* Ileal and/or ileocolonic involvement as demonstrated by most recent endoscopy
* Short CDAI score >150
* Have not received oral or intravenous steroids for >1 month, or with stable dose for >1 month if currently taking
* Stable dose of AZA for >1 month, if currently taking
* Stable dose of anti-TNF inhibitor for >1 month, if currently taking

Exclusion Criteria:

* Pregnant or intend to become pregnant in the next 6 months
* Major abdominal surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
CDAI (Clinical Disease Activity Index) score | 12 weeks
  A statistically significant decrease in CDAI score. The short CDAI score will be utilized for this study. This validated score consists of three subjective, patient-derived measures: (1) number of liquid or soft stools each day for 7 days (2) the sum of seven daily abdominal pain ratings (3) the sum of seven general well-being ratings. The calculation of CDAI score will be as follows: Short CDAI = 44 + (2 × the number of liquid or soft stools each day for 7 days) + [5 × the sum of seven daily abdominal pain ratings (0 = none, 1 = mild, 2 = moderate, 3 = severe)] + [7 × the sum of seven general well-being ratings (0 = generally well, 1 = slightly under par, 2 = poor, 3 = very poor, 4 = terrible). Outcome measures considered to be consistent with benefit from intervention includes either (1) disease remission (CDAI less than 150) or (2) CDAI score reduction of 60 points.
Fecal calprotectin | 12 weeks
  A statistically significant decrease in fecal calprotectin

SECONDARY OUTCOMES:
Morbidity | 12 weeks
  Rates of hospitalization and adverse events

IPD SHARING:
Plan to Share IPD: No